CLINICAL TRIAL: NCT01804972
Title: Efficacy of Patient Centred Information for Vascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mid Western Regional Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Stewart Walsh, Professor Stewart Walsh, Mid Western Regional Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: INFO2013
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Vascular Disease
Keywords: Patient information; Vascular disease; Abdominal aortic aneurysm; Varicose veins; Web based information
MeSH Terms: conditions — Vascular Diseases; Aortic Aneurysm, Abdominal; Varicose Veins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verbal and written infomation (Active Comparator): Verbal and written information:Patients will receive both verbal information and written patient information leaflets
  Interventions: Other: Verbal and written information
- Verbal and electronic information (Experimental): Patient will receive both verbal information and a web address to access patient information electronically
  Interventions: Other: Verbal and electronic information

INTERVENTIONS:
Other: Verbal and written information — Patients will receive verbal information supplied by the attending doctor and also written information in the form of patient information leaflets
  Arms: Verbal and written infomation
Other: Verbal and electronic information — Patients will receive verbal information by the attending doctor and also be provided with a web address to access electronic patient information.
  Arms: Verbal and electronic information

SUMMARY:
This study aims to determine the usefulness of providing patients with web-based electronically accessed patient information when compared to the provision of written information leaflets.

DETAILED DESCRIPTION:
Hospitals and health care institutions attempt to provide information to patients through a variety of media including; written information, web-site based information and more recently through the use of smart phone based applications. Such educational campaigns have financial implications for hospitals and institutions.

The level of knowledge among patients with vascular disease of their pathology and its associated risk factors has been shown to be poor (Lovell et al 2009, Hirsch et al 2007). The optimum tool with which to provide information to patients with vascular disease has not been determined to date.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed abdominal aortic aneurysm, peripheral vascular disease or varicose veins
* Capacity to and willingness to consent to participation in the study
* Adult patients
* In-patient or out-patient status

Exclusion Criteria:

* Previously diagnosed with vascular disease
* Limited capacity or unwilling to consent
* Information already provided by hospital doctor
* Cognitive/intellectual impairment/acquired brain injury/visual impairment
* Qualified medical professionals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Overall improvement in knowledge in a group of patients with vascular disease following the provision of information through verbal, written or electronically based sources. | 6 weeks
  Patients will be randomised to receive either verbal and written information or verbal and electronically based information on their disease specific condition. Knowledge will be assessed through the use of a multi choice questionnaire at baseline prior to the provision of information on their condition and again at follow up 6 weeks later.

SECONDARY OUTCOMES:
Effectiveness of providing electronically based information to the vascular patient population | 6 weeks
  At follow patients will be asked to complete a questionnaire detailing their use of the information provided.
  The following measures will be recorded:
  Did you access the website address provided Y/N
  If Yes, How many times did you access the website (Specify) ____________________
  Did you find the website useful or informative Yes/No/Somewhat
  Did you read the information leaflet provided Y/N
  If Yes, How many times did you read the leaflet (Specify) ______________________
  Did you find the leaflet useful or informative Yes/No/Somewhat

CONTACTS AND LOCATIONS:
Overall Officials: Stewart R Walsh, Principal Investigator — HSE and University of Limerick
Locations (1):
- MidWestern Regional Hospital, Limerick, Limerick, Ireland

REFERENCES:
- [Background] Lovell M, Harris K, Forbes T, Twillman G, Abramson B, Criqui MH, Schroeder P, Mohler ER 3rd, Hirsch AT; Peripheral Arterial Disease Coalition. Peripheral arterial disease: lack of awareness in Canada. Can J Cardiol. 2009 Jan;25(1):39-45. doi: 10.1016/s0828-282x(09)70021-2. PMID 19148341
- [Background] Hirsch AT, Murphy TP, Lovell MB, Twillman G, Treat-Jacobson D, Harwood EM, Mohler ER 3rd, Creager MA, Hobson RW 2nd, Robertson RM, Howard WJ, Schroeder P, Criqui MH; Peripheral Arterial Disease Coalition. Gaps in public knowledge of peripheral arterial disease: the first national PAD public awareness survey. Circulation. 2007 Oct 30;116(18):2086-94. doi: 10.1161/CIRCULATIONAHA.107.725101. Epub 2007 Sep 17. PMID 17875966